CLINICAL TRIAL: NCT03509402
Title: Short vs Long Implants Supporting a Total Fixed Prosthetic Rehabilitation of the Fully Edentulous Mandible. A Multicenter Randomized Controlled Clinical Trial
Brief Title: Short vs Long Dental Implants for the Fixed Rehabilitation of the Fully Edentulous Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Luigi Guida, Full Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEAOUSUN1327012010
Record Dates: First submitted 2018-03-31; First posted 2018-04-26 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Edentulous Jaw
Keywords: short dental implants; full-arch prosthesis
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short implants (Experimental): A full-arch screw-retained mandibular prosthesis with distal cantilevers supported by five interforaminal short implants (ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: 6mm)
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: 6 mm
- Long implants (Active Comparator): A full-arch srew-retained mandibular prosthesis with distal cantilevers supported by five interforaminal short implants (ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: ≥11mm)
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: ≥11mm

INTERVENTIONS:
Device: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: 6 mm — Rehabilitation of the edentulous mandible by a full-arch srew-retained prosthesis with distal cantilevers supported by five interforaminal short implants (ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: 6 mm)
  Arms: Short implants
Device: ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: ≥11mm — Rehabilitation of the edentulous mandible by a full-arch srew-retained prosthesis with distal cantilevers supported by five interforaminal long implants (ASTRA TECH Implant System, OsseoSpeed™ 4.0 S, length: ≥11mm)
  Arms: Long implants

SUMMARY:
The aim of this study is to clinically and radiographically compare the performance of short (6 mm-long) versus long (≥11 mm-long) dental implants placed in the interforaminal region of fully edentulous mandibles, supporting a screw-retained full-arch cantilever bridge.

DETAILED DESCRIPTION:
The use of short dental implants provides undeniable benefits in sites where the reduced available volume would otherwise need bone augmentation procedures and their use has greatly expanded in the recent years. However, well designed clinical trials which provide a sound evidence of their performance and reliability are still lacking to date.

In this post-market, multi-center, open, parallel-group, randomized, controlled clinical trial the investigators aim to to clinically and radiographically compare the performance of short (6 mm-long) versus long (≥11 mm-long) dental implants supporting a mandibular screw-retained full-arch cantilever bridge.

Five 4mm-wide/6mm-long (test) or 4mm-wide/≥11mm-long (control) titanium dental implants (Osseospeed™, ASTRA TECH Implant System™, Dentsply Sirona) are placed in the interforaminal region of fully edentulous mandibles, in non-regenerated sites, with at least 1 mm of peri-implant bone circumferentially.

All products are CE (European Conformity) marked and used within their intended use.

Two-Stage surgery is performed, implants are positioned in healed bone and exposed after 3 months to be connected with the prosthesis.

This is a medium-term follow-up study including evaluations also at 1 and 3 years from the baseline.

Three italian centers participate: Naples (University of Campania "Luigi Vanvitelli"), Naples (AORN "A. Cardarelli"), Catania (Private Office).

The study protocol has been approved by the Institutional Review Board of the University of Campania "Luigi Vanvitelli".

ELIGIBILITY:
Inclusion Criteria:

* total edentulous patients in the lower region since at least 8 months,
* sufficient amount of native bone (no augmentation procedures) in the recipient sites to allow ≥11 mm long and 4 mm wide implant installation (≥1 mm of peri-implant bone circumferentially)
* systemic health
* compliance with good oral hygiene
* informed consent signed.

Exclusion Criteria:

* any disease, medication or drug that could jeopardize healing, osseointegration or treatment outcome,
* untreated caries or periodontitis of the remaining teeth,
* mucosal and bone tissue lesions,
* severe bruxism or other parafunction habits,
* unrealistic aesthetic demands,
* patient taking part to another study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Guida, Prof, Principal Investigator — University of Campania Luigi Vanvitelli

REFERENCES:
- [Background] Albrektsson T, Zarb G, Worthington P, Eriksson AR. The long-term efficacy of currently used dental implants: a review and proposed criteria of success. Int J Oral Maxillofac Implants. 1986 Summer;1(1):11-25. No abstract available. PMID 3527955
- [Background] Nisand D, Renouard F. Short implant in limited bone volume. Periodontol 2000. 2014 Oct;66(1):72-96. doi: 10.1111/prd.12053. PMID 25123762
- [Background] Ekelund JA, Lindquist LW, Carlsson GE, Jemt T. Implant treatment in the edentulous mandible: a prospective study on Branemark system implants over more than 20 years. Int J Prosthodont. 2003 Nov-Dec;16(6):602-8. PMID 14714838
- [Background] Srinivasan M, Vazquez L, Rieder P, Moraguez O, Bernard JP, Belser UC. Survival rates of short (6 mm) micro-rough surface implants: a review of literature and meta-analysis. Clin Oral Implants Res. 2014 May;25(5):539-45. doi: 10.1111/clr.12125. Epub 2013 Feb 18. PMID 23413956
- [Background] Laurell L, Lundgren D. Marginal bone level changes at dental implants after 5 years in function: a meta-analysis. Clin Implant Dent Relat Res. 2011 Mar;13(1):19-28. doi: 10.1111/j.1708-8208.2009.00182.x. PMID 19681932
- [Result] Guida L, Annunziata M, Esposito U, Sirignano M, Torrisi P, Cecchinato D. 6-mm-short and 11-mm-long implants compared in the full-arch rehabilitation of the edentulous mandible: A 3-year multicenter randomized controlled trial. Clin Oral Implants Res. 2020 Jan;31(1):64-73. doi: 10.1111/clr.13547. Epub 2019 Oct 29. PMID 31605405
- [Result] Guida L, Esposito U, Sirignano M, Torrisi P, Annunziata M, Cecchinato D. 6 mm short versus 11 mm long inter-foraminal implants in the full-arch rehabilitation of edentulous non-atrophic mandibles: 5-year results from a multicenter randomized controlled trial. Clin Oral Implants Res. 2023 Feb;34(2):127-136. doi: 10.1111/clr.14024. Epub 2022 Dec 13. PMID 36461704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Implants | Long Implants
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Implants | Long Implants | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6.3) | 61 (8.6) | 63 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 5 | 12 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 15 | 15 | 30
Smoking habit [Count of Participants; unit: Participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level (MBL) Change
Description: Marginal bone level (MBL) is measured as the distance in millimiters calculated on periapical radiographs from the implant neck to the most coronal bone-to-implant contact point at both the mesial and the distal side of each implant. The radiographs will be taken with an X-ray apparatus supplied with a long cone and Rinn's film holders.
Time Frame: 5 years from baseline (prosthetic loading)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Short Implants | Long Implants
Number analyzed (Participants) | 13 | 14
mm | 0.30 (0.31) | 0.40 (0.23)

2. Secondary Outcome: Implant Survival Rate
Description: A surviving implant is defined as an implant in place at the time of the follow-up. Any implant loss shall be assessed as an early loss (implant fails before being osseointegrated) or late loss (after being osseointegrated).
Time Frame: 5 years from baseline (prosthetic loading)
Measure: Number; unit: Implants
Arm/Group | Short Implants | Long Implants
Number analyzed (Participants) | 13 | 14
Implants | 65 | 70

3. Secondary Outcome: Prosthesis Survival
Description: A surviving prosthesis is defined as still in place at the time of the follow-up.
Time Frame: 5 years from baseline (prosthetic loading)
Measure: Number; unit: Prostheses
Arm/Group | Short Implants | Long Implants
Number analyzed (Participants) | 13 | 14
Prostheses | 13 | 14

4. Secondary Outcome: Biological Complications
Description: Peri-implant mucositis and peri-implantitis
Time Frame: 5 years from baseline (prosthetic loading)
Measure: Count of Participants; unit: Participants
Arm/Group | Short Implants | Long Implants
Number analyzed (Participants) | 13 | 14
Participants | 2 | 3

5. Secondary Outcome: Technical Complications
Description: Technical complications are categorized in minor and major complications. The formers require only chair-side repair and include screw loosening and veneer material fracture. The latters require additional laboratory procedures and/or replacement components and include prosthesis or framework fracture, screw fracture, implant fracture, and extended wear requiring veneer renewal.
Time Frame: 5 years from baseline (prosthetic loading)
Measure: Count of Participants; unit: Participants
Arm/Group | Short Implants | Long Implants
Number analyzed (Participants) | 13 | 14
Participants | 7 | 5

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Short Implants | Long Implants
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03509402/Prot_SAP_000.pdf